CLINICAL TRIAL: NCT01875562
Title: A Post-marketing Evaluation of a Compound Traditional Chinese Herbal Medicine, Qishe Pill, on Cervical Radiculopathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Huadong Hospital (Other); Shanghai East Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Shanghai No.1 Hospital (Unknown); Shanghai No.6 Hospital (Unknown); Changhai Hospital (Other)
Responsible Party: Principal Investigator, Cui xuejun, Vice director, Shanghai University of Traditional Chinese Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PME of Qishe
Record Dates: First submitted 2012-12-12; First posted 2013-06-12 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Cervical Radiculopathy
Keywords: Neck pain; Cervical radiculopathy; Qishe Pill; Traditional Chinese Medicine
MeSH Terms: conditions — Radiculopathy; Neck Pain | interventions — qishe

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Qishe Pill (Experimental)
  Interventions: Drug: Qishe Pill

INTERVENTIONS:
Drug: Qishe Pill — Pill, 3.75 g, twice per day, four weeks

SUMMARY:
Neck pain is a common symptom in most patients suffering from cervical radiculopathy. However, some conservative treatments are limited by their modest effectiveness. On the other hand, surgical intervention for cervical disc disorders is indicated when symptoms are refractory to conservative treatments and neurological symptoms are progressive. Many patients use complementary and alternative medicine, including Traditional Chinese Medicine, to address their symptoms. The purpose of the present study is to examine effectiveness and safety of Qishe Pill, a compound traditional Chinese herbal medicine, for neck pain in patients with cervical radiculopathy.

DETAILED DESCRIPTION:
Cervical radiculopathy is a distinct consideration in the evaluation of any patients who have neck pain and may be defined simply as an abnormality of a nerve root which originates in the cervical spine. The initial approach to the management of cervical spondylopathic radiculopathy is nearly the same as that of nonspecific neck or back pain that can be found in most patients. Conservative treatments include non-steroidal anti-inflammatory drugs (NSAIDs), narcotics, muscle relaxants, physical therapy and transcutaneous electrical nerve stimulation (TENS). The main objectives of conservative treatments are to relieve pain, improve function and improve health-related quality of life. However, these treatments for cervical radiculopathy are limited by their modest effectiveness. Surgical treatment for cervical disc disease is indicated when symptoms are refractory to conservative treatments and neurological symptoms are progressive. In terms of pharmacotherapy, there is generally no randomized, placebo-controlled trial available comparing standard nonsurgical treatment. Therefore, care plans should be designed principally based on accumulated experience, the services available locally, and the respective preferences of patients. Treatment plans are developed to alleviate pain, improve function, and prevent recurrences.

As a complementary and alternative medicine (CAM), herbal medicines have the potential to avoid the adverse effects of medications and surgery.According to the basic theory of traditional Chinese medicine (TCM), the obstruction of Qi flow and blood circulation in the neck area caused by pathogenic factors, such as "Feng"(wind), "Han"(cold), "Shi"(dampness), invading the neck induces cervical degenerative disc diseases which are the cause of cervical radiculopathy. According to the four traditional methods of diagnosis -observation, listening, interrogation, and pulse-taking, TCM doctors can analyze the specific pathogenic factors which cause neck pain. Accordingly they can then prescribe herbal formulae based on the effect and the main indications according to the principles of Chinese medicine. Natural substances, including herbal medicines, have been used to promote healing and alleviate neck pain in western countries. Previous studies have demonstrated that some active substances in herbal medicine can promote Qi flow and blood circulation to alleviate pain.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of chronic neck pain since at least 3 months and complaints for a maximum duration of 5 years.
* average pain intensity of the last 7 days more or equal to 25 points measured by a Neck Disability Index.
* intellectual and physical ability to participate in the study. informed consent.
* One positive result of Brachial Plexus Traction Test, Cervical compression test or Cervical distraction test

Exclusion Criteria:

* cervical pain related to malignancy
* cervical pain due to an accident
* inflammatory joint disorders
* previous spine surgery
* protrusion/prolapse of a spinal disk, spondylolisthesis, with radicular symptomatology
* actually doing or planning to do other regular physical exercise during the study with possible positive effects on neck pain - such as swimming, yoga, pilates, tai chi, etc.
* use of pain drugs for other diseases (> 1x/week)
* pregnancy
* severe chronic or acute disease interfering with therapy attendance
* alcohol or substance abuse
* participation in another clinical trial in the last 6 months before study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-10 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
pain severity(measured with a visual analogue scale, VAS) | changes from baseline at 2 weeks
  Operationally, the VAS score display as a horizontal line, 100 mm in length, word descriptors anchored at each end. The patient marks on the line the point that they feel represents their perception of their current pain. The VAS score is then determined by measuring in millimetres from the left hand end of the line to the point that the patient marks.
pain severity(measured with a visual analogue scale, VAS) | changes from baseline at 4 weeks
  Operationally, the VAS score display as a horizontal line, 100 mm in length, word descriptors anchored at each end. The patient marks on the line the point that they feel represents their perception of their current pain. The VAS score is then determined by measuring in millimetres from the left hand end of the line to the point that the patient marks.

SECONDARY OUTCOMES:
SF-36 | changes from baseline at 2 weeks
  a composite of functional status
Neck Disability Index（NDI） | changes from baseline at 2 weeks
  a composite of functional status
SF-36 | changes from baseline at 4 weeks
  a composite of functional status
Neck Disability Index（NDI） | changes from baseline at 4 weeks
  a composite of functional status
Kidney function test | changes from baseline at 4 weeks
Liver function test | changes from baseline at 4 weeks
ECG | changes from baseline at 4 weeks
Occult Blood | changes from baseline at 4 weeks
Urine routine | changes from baseline at 4 weeks
Blood routine | changes from baseline at 4 weeks
Number of participants with Concomitant medication | 4 weeks
Number of participants with Adverse Events | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, Dr, Principal Investigator — Longhua Hospital
Locations (1):
- Longhua Hospital, Shanghai University of TCM, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Cui XJ, Sun YL, Zhang CQ, Wu T, Tan J, Zhu ZA, Chen YQ, Wang QG, Li M, Wang YJ. Post-Marketing Surveillance of Qishe Pill () Use for Management of Neck Pain in a Chinese Patient Cohort to Determine its Safety, Tolerability and Effectiveness. Chin J Integr Med. 2021 Jun;27(6):408-416. doi: 10.1007/s11655-021-2868-x. Epub 2021 Apr 21. PMID 33881718